CLINICAL TRIAL: NCT06711263
Title: Role of Herbal Based Mouthwashes in Plaque Control. a Randomized Clinical Control Trial
Brief Title: Role of Herbal Based Mouthwashes in Plaque Control
Acronym: mouthwash
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Dr, Ajman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Ajman Herbal mouthwash 2425
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Plaque Induced Gingival Disease
Keywords: plaque; gingival bleeding; resveratrol; miswak; tea tree oil; chlorhexidine
MeSH Terms: conditions — Plaque, Amyloid; Gingival Hemorrhage | interventions — Chlorhexidine; Tea Tree Oil

STUDY DESIGN:
Intervention Model Description: In the Initial Visit-Baseline, and subsequent visits, participants will be called in the morning. Morning hours will be chosen for examination, as it will reduce the risk of bias and also help in quantifying results. plaque and gingival scores will be recorded and the First herbal mouthwashes will be given, participants will also be provided new tooth-brushes (Oral B-soft).
Who Masked: Participant
Masking Description: participants are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- chlorhexidine (Experimental): Mouthwash will be used for these participants
  Interventions: Other: Mouthwash Product
- Tea tree oil (Active Comparator): Participants will use the mouthwash and plaque and gingival bleeding indice will be recorded at baseline, after 2 weeks and after 4 weeks
  Interventions: Other: Mouthwash Product
- Reseverotriol (Active Comparator): Participants will use the mouthwash and plaque and gingival bleeding indice will be recorded at baseline, after 2 weeks and after 4 weeks
  Interventions: Other: Mouthwash Product
- Miswak (Active Comparator): Participants will use the mouthwash and plaque and gingival bleeding indice will be recorded at baseline, after 2 weeks and after 4 weeks
  Interventions: Other: Mouthwash Product

INTERVENTIONS:
Other: Mouthwash Product — * In the Initial Visit-Baseline, and subsequent visits, participants will be called in the morning. Morning hours will be chosen for examination, as it will reduce the risk of bias and also help in quantifying results. plaque and gingival scores will be recorded and the First herbal mouthwashes will be given, participants will also be provided new tooth-brushes (Oral B-soft).
  * They will be asked to follow their routine oral hygiene habits. They will be asked to come back after 2 weeks for plaque and gingival bleeding scores recording for the second visit and again after 2weeks post the second visit for the third and final visit to record their plaque and gingival bleeding scores.
  Other Names: chlorhexidine; resverotriol; miswak; tea tree oil

SUMMARY:
Herbal medicine has been used for thousands of years. Traditional herbal medicine is used by an estimated 80% of the world's population for primary health care. Herbal treatments have gained popularity as a dietary supplement for illness prevention and as an alternative/complementary therapy in recent years. Herbal remedies come in a wide variety of forms and can be found on the market all over the world.

DETAILED DESCRIPTION:
Herbal mouthwashes have been increasingly popular over time. Ethnomedicines are the term used to describe them. Various substances have been tested, with phytopharmacological analyses yielding contradictory results. Many previous studies had tested the antiplaque efficiency of one herbal mouthwash with contradicting results, other studies have tested the Antiplaque efficiency of chlorhexidine, tea tree oil and Miswak, some studies had given positive outcomes and benefits of Miswak on the gingiva and others when comparing between the efficacy of Miswak over chlorhexidine mouth wash in dental practice provided results favouring both these mouthwashes.

In our proposed study we will compare the antiplaque efficiency of three herbal kinds of mouthwash, Miswak, tea tree oil and Resveratrol mouthwash. Plaque and gingival bleeding scores will be taken before the study from 6 different teeth and retaken after 2 weeks and four weeks respectively the use of the mouthwash. This study is single-blinded. Antiplaque and gingival bleeding scores from the three mouthwashes will be recorded over a period of a month and statistical analysis will be performed

ELIGIBILITY:
Inclusion Criteria:

* Patients who are medically fit
* Patients with gingival inflammation not progressed into periodontitis (AAP classification
* Patients between the age of 18-60 years

Exclusion Criteria:

* Patients who are medically compromised
* Patient who have undergone a periodontal therapy for the past 3 months
* Patients who are healthy but have been using herbal mouthwashes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
plaque score | From Baseline-pre-intervention to the end of treatment at 4 weeks
  To assess the plaque score

SECONDARY OUTCOMES:
gingival bleeding score | from pre-intervention to the end of the treatment at 4 weeks
  To assess gingival bledding score

IPD SHARING:
Plan to Share IPD: No